CLINICAL TRIAL: NCT03450824
Title: Research on the Relationship Between Constitutional Varus Knee and Patellofemoral Pain
Brief Title: Relationship Between Constitutional Varus Knee and Patellofemoral Pain
Status: Terminated | Type: Observational
Why Stopped: Because not enough volunteers were recruited.
Sponsor: 113th Hospital of Chinese People's Liberation Army (Other)
Collaborators: Air Force Military Medical University, China (Other)
Responsible Party: Sponsor
Other Study IDs: 113YY-LUNLI-2018002
Record Dates: First submitted 2018-02-23; First posted 2018-03-01 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Patellofemoral Pain Syndrome
Keywords: Patellofemoral Pain Syndrome; Anterior Knee Pain; Knee Varus
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- The study group: The participants with patellofemoral pain.
  Interventions: Other: No intervention
- The control group: The participants without patellofemoral pain.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — The standardized standing whole-lower-extremity radiographs, the knee lateral view and skyline view of the participants will be taken.

SUMMARY:
This study aims to research on the relationship between constitutional varus knee and patellofemoral pain. The standardized standing whole-lower-extremity radiographs, the knee lateral view and skyline view of the participants will be taken. The hip-knee-ankle angle will be obtained from the radiographs. According to the hip-knee-ankle angle, the knees will be labelled knee varus or knee nonvarus. The knee varus incidences of the two groups will be determined and compared.

DETAILED DESCRIPTION:
The patellofemoral joint will be assessed in the skyline view and lateral view. The hip-knee-ankle angle will be obtained from the standing whole-lower-extremity radiographs. According to the hip-knee-ankle angle, the knees will be labelled knee varus or knee nonvarus. The knee varus incidences of the two groups will be determined and compared. It is hypothesized that constitutional varus knee is a risk factor for patellofemoral pain.

ELIGIBILITY:
Inclusion Criteria:

* Patellofemoral pain during physical activities such as running, jumping, squatting, and going up or down stairs for at least 4 weeks.
* The onset of pain is required to be atraumatic in nature.
* Exhibit two of the following clinical criteria on assessment: pain on direct compression of the patella against the femoral condyles with the knee in full extension, tenderness of the posterior surface of the patell on palpation, pain on resisted knee extension, and pain with isometric quadriceps muscle contraction against suprapatellar resistance with the knee in 15° of flexion.
* Negative findings in the examination of knee ligaments, menisci, bursae, synovial plicae, Hoffa's fat pad, iliotibial band, and the hamstring, quadriceps, and patellar tendons and their insertions.

Exclusion Criteria:

* With patellofemoral instability, or With other knee diagnoses.
* Any previous surgery or severe trauma in the affected limb.
* Inflammatory joint disease or tumors in the affected limb.

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Military personnel. Running at least 10 km per week for at least 3 months.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2018-03-23 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-06-15 (Actual)

PRIMARY OUTCOMES:
The hip-knee-ankle angle | 1 day
  The HKA angle was determined by measuring the angle between the mechanical axis of the femur and the mechanical axis of the tibia.

SECONDARY OUTCOMES:
Patellar alignment | 1 day
  The lateral displacement of the patella was defined as the proportion of the distance from the lateral edge of the patella to a line drawn perpendicular to a line passing along the most anterior margin of the medial and lateral trochlear facets, by the length of the maximum width of the patella. The tilting angle of the patella was defined as the angle formed by a line joining the maximum width of the patella and a line passing along the most anterior margin of the medial and lateral trochlear facets.
The width of of the patellofemoral joint space | 1 day
  The width of the joint space at the mid-point of the medial and lateral patellofemoral joint is measured on the skyline view.
Trochlear morphology | 1 day
  The sulcus angle was defined as the angle between the medial and lateral trochlear facets. The vertex of the angle was the deepest portion of the trochlea.
Patellar height | 1 day
  The Insall-Salvati ratio is the ratio between the length of the patellar tendon and the superior-inferior length of the patella.

CONTACTS AND LOCATIONS:
Overall Officials: Qingsheng Zhu, MD, Study Director — Department of orthopaedics, Xijing hospital, Fourth Military Medical University, Xi'an, China
Locations (1):
- Orthopaedics clinic, No.113 Hospital of Chinese People's Liberation Army, Ningbo, Zhejiang, China